CLINICAL TRIAL: NCT05029804
Title: The Effect of Walking Exercise Training Based on the Theoretical Model on Adherence to Disease Management and Metabolic Control in Type 2 Diabetes Patients: A Clinical Randomized Controlled Study
Brief Title: Effect of Walking Exercise Training on Adherence to Disease Management and Metabolic Control in Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gulengul Mermer, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Type2DiabetesEge
Record Dates: First submitted 2021-08-19; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2; Exercise; Walking Pneumonia; Diabetes
Keywords: Diabetes Mellitus, Type 2; Transtheoritical Model; Walking; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Pneumonia, Mycoplasma; Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After the initial assessment, patients in this group will be educated by the researcher on walking exercise by using the transtheoritical model. The data will be collected from the patients in the experimental group at baseline, 1st, 3rd, and 6th months of the programme.
  The data will be collected by using Exercise Stages of Change Questionnaire, Exercise Processes of Change Scale, Pedometer, Patient Compliance in Type 2 Diabetes Mellitus Treatment Scale, and patient identification that includes five domain. These domains include questions about the patients' sociodemographic characteristics, habits, knowledge of diabetes and its treatment, exercise status, and the evaluation of the metabolic control variables.
  Interventions: Other: Education
- Control (No Intervention): No intervention will be applied to this group. The data will be collected from the patients in the control group at baseline, 1st, 3rd, and 6th months.
  The data will be collected by using Exercise Stages of Change Questionnaire, Exercise Processes of Change Scale, Pedometer, Patient Compliance in Type 2 Diabetes Mellitus Treatment Scale, and patient identification that includes five domain. These domains included questions about the patients' sociodemographic characteristics, habits, knowledge of diabetes and its treatment, exercise status, and the evaluation of the metabolic control variables.

INTERVENTIONS:
Other: Education — This intervention will be applied to the patients in the experimental group. The education will be provided by the researcher and based on the transtheoritical model. Printed materials and PowerPoint presentations will be used for the education and the education will be conducted in a face-to-face session with each participant (10 weeks).
  Arms: Intervention Group

SUMMARY:
This study aims to determine the effects of a transtheoretical model-based walking exercise training and disease management and metabolic control in patients with type 2 diabetes. This randomized controlled trial will be conducted as a pre-test and post-test experiment with 30 intervention and 30 control individuals. The intervention group will receive the transtheoretical model-based exercise training. The intervention group will be followed-up for 6 months (from 0 to 6 months) to determine the patients' behavioral changes after the training will be completed.

DETAILED DESCRIPTION:
This study aims to determine the effects of a transtheoretical model-based walking exercise training and disease management and metabolic control in patients with type 2 diabetes. This randomized controlled trial will be conducted as a pre-test and post-test experimental model with 30 intervention and 30 control individuals. The intervention group will receive the transtheoretical model-based exercise training. Data will be collected using patient a identification form, Patient Compliance Scale to the Treatment of Type 2 Diabetes Mellitus, transtheoretical model scales, pedometer and metabolic outcomes. Data will be analyzed by using Chi square, two-way ANOVA to determine the difference between two or more independent/dependent groups and Spearman's correlation to determine the relationship between two groups.

ELIGIBILITY:
Inclusion Criteria:

Patients who diagnosed with type 2 diabetes at least 6 months. Received insulin and/or oral antidiabetic treatment, literate, and having no communication problems, between the ages of 18 and 65, whose arterial blood pressure is in range of systolic ≤ 160mmHg and diastolic ≤ 100mmHg, who had HbA1c between 7-9 % will be included in the study. The patients who agree to participate in the study (voluntarily) and who have no objection to exercising with cardiology consultation will be included in the study.

Exclusion Criteria:

Participants with diabetes-related (severe) complications and diabetic foot, pregnancy, diagnosed with cancer, having physical and mental problems that prevent walking will be excluded from the study. HA1C over 9 - despite the treatment (will be referred to the doctor for treatment change). Patients with blood sugar above 300 - despite treatment (will be referred to their doctor for a change in treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic Parameters 1 | The change in 6 months from baseline
  Fasting Blood Glucose (mg/dL), the fasting blood glucose will be assessed by taking blood sample from the patients.sample from the patients.
Metabolic Parameters 2 | The change in 6 months from baseline
  HbA1c (both % and mmol/mol), the HbA1c will be assessed by taking blood sample from the patients.
Metabolic Parameters 3 | The change in 6 months from baseline
  Total cholesterol (mg/dL), the total cholesterol will be assessed by taking blood sample from the patients.
Metabolic Parameters 4 | The change in 6 months from baseline
  Creatinine (mg/dL), the creatinine will be assessed by taking blood sample from the patients.
Exercise Stages of Change Questionnaire | The change in 6 months from baseline
  Prochaska et al. (1992) studied how people change. Marcus et al. developed a structured questionnaire to measure the stages of exercise changes. Ay and Temel (2015) adapted the questionnaire to Turkish society. The scale consists of five questions about the patient's stage of change (prethinking, thinking, preparation, taking action, and maintenance). In the pre-thinking stage, the patients do not plan to start exercise now or during the next 6 months. The patients in the thinking stage do not make an effort to exercise actively, but intend to start in the next 6 months. The patients in the preparation stage intend to start exercising regularly in the next 30 days. The patients in the taking action stage have started exercising within the last 6 months. The patients in the maintenance stage continue to change over the course of the action, exercise more than 6 months and are confident and determined not to return to previous behavior.
Exercise Processes of Change Scale | The change in 6 months from baseline
  The exercise processes of change scale was developed by Marcus et al. and adapted to Turkish society by Ay and Temel. Exercise processes of change is based on a 5-point Likert type scale and consists of 28 items. The maximum score that a patient can obtain on the scale is 140, the minimum score is 28. The scale consists of 10 sub-dimensions and two main processes (behavioral and cognitive). Behavioral processes are opposition, helping relationships, empowerment management, self-emancipation and stimulus control. Cognitive processes are increased awareness, dramatic help, environmental reassessment, self reassessment, social independence. The higher the scale score is indicates a higher success of the change. In this study, the general Cronbach alpha reliability coefficient of the scale was determined as 0.96 (behavioral process = 0.94 and cognitive process = 0.93).
Patient Compliance in Type 2 Diabetes Mellitus Treatment Scale | The change in 6 months from baseline
  This scale consists of 30 questions and a five-point Likert type rating is used. There are 13 positive and 17 negative items in the scale. Scoring ranges from 1 to 5 for positive items, and reverse scoring ranges from 5 to 1 for negative items. The highest score obtained from the scale is 150, the lowest score is 30. 30-54 points from the scale indicates "good adherence to treatment", 55-125 points "medium adherence to treatment", and 126-150 points indicate that the patient's adherence to treatment is poor. The scale was developed by Demirtaş and Albayrak for use in Turkish society. Cronbach's alpha value was found to be 0.77.
Pedometer | The change in 6 months from baseline
  A pedometer is a portable, small, inexpensive, and objective tool used to measure the number of steps. The pedometer includes a mechanical motion sensitive sensor that detects movements during walking. To prevent diseases and encourage healthy lifestyles, 150 minutes exercise and 10,000 steps per day are recommended. The researcher will provide participants with Omron brand HJ-320-E model pedometers to record 7days of activity data. These records were used to calculate the average number of steps per day.

CONTACTS AND LOCATIONS:
Overall Officials: Gulengul Mermer, Study Director — Ege Uninersity

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data to other researchers